CLINICAL TRIAL: NCT02917668
Title: Evaluation of the Risk of Hyperoxia-induced Hypercapnia in Obese Patients in a Cardiac Surgery Postoperative Setting
Brief Title: Evaluation of the Risk of Hyperoxia-induced Hypercapnia in Obese Cardiac Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, François Lellouche, MD, PhD, Laval University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 21366
Record Dates: First submitted 2016-09-25; First posted 2016-09-28 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Obesity; Hyperoxia; Hypercapnia
Keywords: Obesity; Hyperoxia; Hypercapnia; Postoperative complications; Cardiac surgical procedures
MeSH Terms: conditions — Obesity; Hyperoxia; Hypercapnia; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): 15 patients who will receive usual care for 30 minutes and then switch to FreeO2 for another 30 minutes
  Interventions: Other: FreeO2; Other: Usual care
- Group B (Active Comparator): 15 patients who will be oxygenated by FreeO2 for 30 minutes and then switch to usual care for another 30 minutes
  Interventions: Other: FreeO2; Other: Usual care

INTERVENTIONS:
Other: FreeO2 — Oxygen delivery automatically titrated by a closed-loop system that adjusts the oxygen flow based on the patient's real-time SpO2 and a programed SpO2 target of 90 %
Other: Usual care — Oxygen delivery manually titrated by the nursing staff for a SpO2 target of > or = 95 %

SUMMARY:
This study aims to evaluate the risk of hyperoxia-induced hypercapnia in post-op obese cardiac surgery patients. It will compare two oxygenation modes in terms of their effect on the arterial partial pressure of carbon dioxide (PaCO2) : manual titration of oxygen delivery for a peripheral oxygen saturation (SpO2) target of > or = 95 % versus automatic titration by a closed-loop system for a SpO2 target of 90%. 15 post-op obese cardiac surgery patients will be recruited and each will receive both interventions (cross-over design). The main outcome will be the PaCO2, which will be compared after each study period. The research hypothesis is that the usual SpO2 target of > or = 95 % is associated with a greater PaCO2 compared with a lesser SpO2 target of 90%.

DETAILED DESCRIPTION:
This study aims to evaluate the risk of hyperoxia-induced hypercapnia in post-op obese cardiac surgery patients.

The investigators will compare two oxygenation modes in terms of their effect on PaCO2 : a SpO2 target of > or = 95 % achieved with manual titration (usual practice) and a more conservative SpO2 target of 90 % achieved with automatic titration by a closed-loop system (FreeO2).

The choice of a SpO2 target of 90 % is consistent with recent guidelines issued by the British Thoracic Society and the Thoracic Society of Australia and New Zealand, which both recommend a SpO2 target of 88-92 % for morbidly obese patients (BMI > 40 kg/m2).

FreeO2 is a closed-loop oxygen delivery system which adjusts the oxygen flow according to the patient's real-time SpO2 and a target programed by the physician. The system also records data on heart rate, respiratory rate and SpO2. Its safety and efficacy have been tested in healthy subjects as well as in patients suffering from COPD or acute respiratory distress in the emergency room, with promising results.

The research hypothesis is that the usual SpO2 target of > or = 95 % is associated with a greater PaCO2 compared with a lesser SpO2 target of 90%.

30 obese patients will be recruited* at the Institut universitaire de cardiologie et de pneumologie de Québec. A written consent from the patient will be obtained the day before the surgery. The protocol has been submitted to and approved by the establishment's ethics committee.

The study will compare the effect of two different oxygenation modes on the patients' PaCO2 immediately after extubation :

FreeO2 mode : oxygen delivered by nasal cannula or Venturi mask (if flow > 5L/min during > 5 minutes), automatically titrated for a SpO2 of 90 +/- 2 %

Usual mode : oxygen delivered by Venturi mask, manually titrated for a SpO2 superior or equal to 95 % (the local protocol is to deliver a post-extubation FiO2 which is 10 % superior to the pre-extubation FiO2)

Patients meeting all of the eligibility criteria will be randomized in the postoperative period. After extubation, they will receive oxygen for 30 minutes according to FreeO2 mode or the usual mode, depending on randomization. After 30 minutes, a first arterial blood gas will be obtained through their arterial cannula. Next, they will be oxygenated according to the second oxygenation mode for another 30 minutes, after which a second arterial blood gas will be obtained. Each patient will thus act as his own control (cross-over design).

When patients will be oxygenated according to the usual mode, FreeO2 will be in recording mode, but will not be delivering any oxygen.

The study will last 1h for each patient, and will have to begin within 30 minutes after extubation. A member of the research team will be at the patient's bedside for the whole data collecting period.

Complete data collection should be achieved within 12 months.

Demographic data (age, sex, weight, height and BMI) will be collected upon study entering as well as pre-operative room air PCO2 on capillary blood gas, type of surgery (number of bypass grafts, extracorporal circulation time), opiates dosage per-op and post-op, and pre-op left ventricular ejection fraction and renal function. FreeO2 will be recording respiratory rate, heart rate and SpO2 for the whole study duration. The respiratory rate will also be recorded manually and on the monitor. When patients will be receiving oxygen from FreeO2, the system will record the delivered flow ; with the usual mode, the staff will record the delivered FiO2. At the end of each intervention, hemodynamic measures will be taken : systolic, diastolic and median arterial blood pressure, systolic, diastolic and median pulmonary artery pressure and amine level.

*Initially, 15 patients were supposed to be included. After inclusion of those 15 patients, statistical analyses showed a lack of statistical power and a possibly significant difference in PaCO2, but only in half the patients. We thus submitted a protocol amendment to our institution's ethics committee to enlarge the sample size to 30 patients, which was accepted on July 13th, 2017.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 kg/m2
* SpO2 > or = 95 % before extubation
* Procedure : coronary artery bypass

Exclusion Criteria:

* Comorbidities : chronic obstructive pulmonary disease, cystic fibrosis, restrictive syndrome not associated with obesity (pulmonary fibrosis, neuromuscular junction disease, etc.)
* Obstructive sleep apnea requiring a positive-pressure mask in the posteoperative period
* FreeO2 device unavailable
* Inclusion in another study that does not permit dual inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09; Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Difference in PaCO2 | At 30 minutes (first intervention) and at 1h (second intervention)
  Difference in end-of-period PaCO2 on arterial blood gas

SECONDARY OUTCOMES:
Difference in pH | At 30 minutes (first intervention) and at 1h (second intervention)
  Difference in end-of-period pH on arterial blood gas
Difference in PaO2 | At 30 minutes (first intervention) and at 1h (second intervention)
  Difference in end-of-period PaO2 on arterial blood gas
Difference in percentage of time spent in hypoxemia (SpO2 < 88%) | In the first 30 minutes (first intervention) and between 30 min and 1h (second intervention)
  Difference in percentage of time spent in hypoxemia (SpO2 < 88%) between periods
Difference in percentage of time spent in severe hypoxemia (SpO2 < 85 %) | In the first 30 minutes (first intervention) and between 30 min and 1h (second intervention)
  Difference in percentage of time spent in severe hypoxemia (SpO2 < 85 %) between periods
Difference in percentage of time spent in hyperoxemia (SpO2 > 96 %) | In the first 30 minutes (first intervention) and between 30 min and 1h (second intervention)
  Difference in percentage of time spent in hyperoxemia (SpO2 > 96 %) between periods
Difference in respiratory rate (manual and monitor) | At 0, 10, 20, 30, 40, 50 and 60 minutes
  Difference in respiratory rate (manual, monitor, FreeO2) between periods for each measuring technique (manual and monitor)
Difference in mean heart rate | In the first 30 minutes and between 30 and 60 minutes
  Difference in mean heart rate, recorded continuously by FreeO2, between periods
Difference in arterial blood pressure | At 0, 10, 20, 30, 40, 50 and 60 minutes
  Difference in arterial blood pressure (systolic, diastolic and mean) between periods
Difference in pulmonary artery pressure | At 0, 10, 20, 30, 40, 50 and 60 minutes
  Difference in pulmonary artery pressure (systolic, diastolic and mean) between periods
Difference in vasopressor dosage | At 0, 10, 20, 30, 40, 50 and 60 minutes
  Difference in vasopressor dosagel at different times between periods
Difference in body temperature | At 0, 10, 20, 30, 40, 50 and 60 minutes
  Difference in body temperature at different times between periods

CONTACTS AND LOCATIONS:
Overall Officials: François Lellouche, MD, PhD, Principal Investigator — Laval University
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The investigators would like to publish our results in scientific magazine and/or present them in a Conference.

REFERENCES:
- [Background] Beasley R, Chien J, Douglas J, Eastlake L, Farah C, King G, Moore R, Pilcher J, Richards M, Smith S, Walters H. Thoracic Society of Australia and New Zealand oxygen guidelines for acute oxygen use in adults: 'Swimming between the flags'. Respirology. 2015 Nov;20(8):1182-91. doi: 10.1111/resp.12620. PMID 26486092
- [Background] O'Driscoll BR, Howard LS, Davison AG; British Thoracic Society. BTS guideline for emergency oxygen use in adult patients. Thorax. 2008 Oct;63 Suppl 6:vi1-68. doi: 10.1136/thx.2008.102947. No abstract available. PMID 18838559
- [Background] Lellouche F, L'her E. Automated oxygen flow titration to maintain constant oxygenation. Respir Care. 2012 Aug;57(8):1254-62. doi: 10.4187/respcare.01343. Epub 2012 Feb 17. PMID 22348812
- [Derived] Denault MH, Ruel C, Simon M, Bouchard PA, Simard S, Lellouche F. Evaluation of hyperoxia-induced hypercapnia in obese patients after cardiac surgery: a randomized crossover comparison of conservative and liberal oxygen administration. Can J Anaesth. 2020 Feb;67(2):194-202. doi: 10.1007/s12630-019-01500-x. Epub 2019 Oct 24. PMID 31650500

DOCUMENTS (1):
  • Study Protocol (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT02917668/Prot_000.pdf